CLINICAL TRIAL: NCT04173052
Title: Sperms Activation by Direct Electrical Shocks on Testis in Infertile Males
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Hashim Talib Hashim, Principal Investigator, University of Baghdad
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A12345
Record Dates: First submitted 2019-11-18; First posted 2019-11-21 (Actual); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Infertility
Keywords: Infertility; Electrical shock; sperms activation; Semen Analysis
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Infertile Males (Experimental): It represents the participants, all the participants in the study are infertile.
  Interventions: Device: Testis' shocker

INTERVENTIONS:
Device: Testis' shocker — The device gives electrical shock ranged (1-5) milliAmpere designed to fit the testis shape for the males.
  Other Names: JT®

SUMMARY:
Background :

Up to 15 percent of couples are infertile. In up to half of these couples, male infertility plays a role. Male infertility is due to low sperm production, abnormal sperm function or blockages that prevent the delivery of sperm. Illnesses, injuries, chronic health problems, lifestyle choices and other factors can play a role in causing male infertility.

Methodology :

It is an interventional trial that involved 45 participants with infertility (Oligospermia, Hypospermia, Asthenozoospermia and Necrozoospermia). All the participants underwent a semen analysis for his semen count, volume and motility for a sample taken by masturbation. Then I gave each one of the participants a small device. This device gives an electrical shock up to 5 milliamps. I told each one independently to use this device properly on his testis every day and come for follow up checking every month.

After the fourth months, I made the final checkup for everyone and records my data and make a comparison between (before and after) semen analysis.

DETAILED DESCRIPTION:
Introduction :

Up to 15 percent of couples are infertile. (1) This means they aren't able to conceive a child even though they've had frequent, unprotected sexual intercourse for a year or longer. In up to half of these couples, male infertility plays a role. Male infertility is due to low sperm production, abnormal sperm function or blockages that prevent the delivery of sperm. Illnesses, injuries, chronic health problems, lifestyle choices and other factors can play a role in causing male infertility. (2,3) Not being able to conceive a child can be stressful and frustrating, but a number of male infertility treatments are available. The consequences of infertility are manifold and can include societal repercussions and personal suffering. Advances in assisted reproductive technologies, such as IVF, can offer hope to many couples where treatment is available, although barriers exist in terms of medical coverage and affordability. (4) Electrical shocks are applied in many fields to treat many diseases especially in psychiatry and mental disorders. Despite its hazards but it can be useful within range of current (Up to 5 milliamps). In 1 milliamp can cause just a faint tingle, this tingle increases as the amount of current increasing until it causes a little pain with 5 milliamps. (5,6,7)

Methodology:

It is an interventional trial that involved 45 participants with infertility (Oligospermia, Hypospermia, Asthenozoospermia and Necrozoospermia) aged (25 - 45 years) and all of them were married. 5 participants were excluded because they have Aspermia or Azoospermia. After clarifying the purpose and the mechanism of the study to the participants, all of them signed a written consent for each one to confirm his agreement to participate in addition to the little risks that can be brought as result of the trial if there is. The investigator applied a semen analysis at a licensed laboratory in Dhi Qar, Nassiryah city in the north of Iraq by many Laboratory assistances under the supervision of an infertility specialist. All the participants underwent a semen analysis for his semen count, volume and motility for a sample taken by masturbation. After choosing my participants and selecting their conditions. Then The investigator gave each one of the participants a small device (Created by an electrical engineer from Dhi Qar Engineering College). This device gives an electrical shock up to 5 milliamps. The investigator told each one independently to use this device properly on his testis every day and come for follow up checking every month as follow:

1. The first month: 1 milliamp for the first 15 days and 2 milliamps for the second 15 days.
2. The second month: 3 milliamps.
3. The third month: 4 milliamps. This process continued for four months (1st June - 25th September, 2019) with regular follow up by semen analysis. After the fourth months, The investigator made the final checkup for everyone and records my data and make a comparison between (before and after) semen analysis and the follow up semen analysis using Statistical Package for the Social Science (SPSS) version 24.

Discussion:

When The investigator compared between the fourth semen analysis results, The investigator found a clear change and improvement in seminal motility, volume and count. This can be used in treating patients with infertility by applying a small amount of current on the testis from outside (taking in consideration the skin and tissues) which can improve the movement and power of the sperms gradually and it is also painless.

It is also can be used before intercourse time for those who are very hurry to fertilize an ovum so their chance of getting an embryo will increase. This device can be produced so any person with infertility (Oligospermia, Hypospermia, Asthenozoospermia and Necrozoospermia) can get one and use it with instructions to make his sperms more powerful to fertilize an ovum.

ELIGIBILITY:
Inclusion Criteria:

* Males with (Oligospermia, Hypospermia, Asthenozoospermia and Necrozoospermia)

Exclusion Criteria:

* Males with (Aspermia or Azoospermia)

Ages: 25 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09-20 (Actual); Study Completion 2019-09-25 (Actual)

PRIMARY OUTCOMES:
Sperms movement | 3 months
  Monitoring the changes that could occur in the motility of the sperms for each participant and record that.
Sperms' number | 3 months
  Monitoring the changes that could occur in the numbers of the sperms for each participant and record that.

CONTACTS AND LOCATIONS:
Overall Officials: Hashim T Hashim, MD, Principal Investigator — University of Baghdad / College of Medicine
Locations (1):
- Al- Nassiryah Laboratory's, Baghdad, Iraq

REFERENCES:
- [Derived] Hashim HT, Varney J, Qais Z, Reda A, Qaderi S, Chowdhury NS, Murry K, Shah J, Alhaideri A, Ahmad S, Hashim AT, Rehman R, Ahmed N, Al-Jorani MS, Skuk M, Abdalhusain M, Khalafalla K. Direct and Gradual Electrical Testicular Shocks Stimulate Spermatogenesis and Activate Sperms in Infertile Men: A Randomized Controlled Trial. Am J Mens Health. 2024 Nov-Dec;18(6):15579883241296881. doi: 10.1177/15579883241296881. PMID 39601214